CLINICAL TRIAL: NCT01974232
Title: A Retrospective Chart Review of Thirty Three Children Who Have Received Clinical Treatment With Either Romiplostim or Eltrombopag From 2009-2013
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Other Study IDs: 1310014390
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia (ITP), Thrombopoietin (TPO) agents, children, romiplostim and eltrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Jacobs syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Romiplostim group
- Eltrombopag group

SUMMARY:
This is a retrospective analysis of children (≤21years old) who received clinical treatment with either Romiplostim or Eltrombopag at 2 medical centers from 2009-2013. The children included in this study were from Weill Medical College of Cornell University, New York, New York and Children's Hospital Orange County, Orange, California

ELIGIBILITY:
Inclusion Criteria:

1. All patients in this study had received prior treatments before the start of TPO treatment including corticosteroids, IVIG, IV anti-D, and/or Rituximab.

Exclusion Criteria:

1. Children who do not have ITP

Ages: 19 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients eligible for this study included both males and females ≤ 21 years old (actual range 19 months - 19 years) with persistent/chronic ITP lasting >6 months and were diagnosed according to the clinical practice guidelines from the American Society of Hematology.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Platelet count greater than or = to 50,000 | on two consecutive weeks

SECONDARY OUTCOMES:
An increase in platelets greater than or = to 20,000 over baseline. | On two consecutive weeks

OTHER OUTCOMES:
Percentage of weeks with platelet counts greater than or = to 50,000 independent of rescue therapy. | For Rescue therapy is defined as receiving Intravenous Immunoglobulin (IVIG) increased dose steroids or platelet transfusions . When given this resulted in exclusion of platelet counts for 2 full weeks after indication of rescue therapy ..

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No